CLINICAL TRIAL: NCT06664346
Title: Exploring the Potential of a Cognitive Mindfulness Intervention Using Virtual Reality to Address Academic Procrastination and Academic Engagement in a London University: A Brief Waitlist Pilot Randomised Controlled Study
Brief Title: Cognitive Mindfulness Intervention Using Virtual Reality to Address Academic Procrastination and Academic Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Metropolitan University (Other)
Responsible Party: Principal Investigator, Samantha Banbury, Principal Investigator, London Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: London University
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Procrastination
Keywords: Academic procrastination; Academic engagement; Immersive cognitive mindfulness; Perceived academic stress

STUDY DESIGN:
Intervention Model Description: Participants were randomised to an active or delayed group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Immersive virtual reality mindfulness intervention software including focus and calm along with mindfulness breathing exercises
  Interventions: Behavioral: Immersive virtual reality mindfulness
- Delayed group (Active Comparator): Immersive virtual reality mindfulness intervention software including focus and calm along with mindfulness breathing exercises
  Interventions: Behavioral: Immersive virtual reality mindfulness

INTERVENTIONS:
Behavioral: Immersive virtual reality mindfulness — Immersive virtual reality mindfulness

SUMMARY:
The study aimed to establish the effectiveness of an immersive mindfulness virtual reality intervention using mindfulness software for students experiencing academic procrastination.

It was hypothesised that post immersive virtual reality mindfulness intervention would result in higher academic self efficacy, lower academic procrastination, and perceived academic stress levels with higher academic engagement. It was further hypothesised that in physiological responses, the pulse rate would be lower post-intervention per session and an overall reduction in pulse rate post intervention.

DETAILED DESCRIPTION:
Virtual reality is a powerful tool that creates a simulated virtual environment, offering immersive and non immersive options. The latter, which refers to the absence of a headset, is controlled by a computer screen using a keyboard and mouse. An immersive example is Meta Quest, a head mounted display that is more economically feasible and accessible. The use of virtual reality in pedagogy, while still in its early stages, is gaining popularity in various educational settings. The potential of virtual reality technology in mindfulness is an exciting prospect that warrants further exploration, offering a new and innovative approach to addressing academic procrastination and engagement. Research has identified the benefits of mindfulness for procrastination among students; however, minimal clinical trials are looking at how immersive virtual reality using mindfulness can support procrastination among students.

The study's design compared the differences in cognitive mindfulness, academic stress, academic procrastination, self efficacy and academic engagement measured with the delayed and active groups at weeks 0, 4, and 12. A waitlist randomised controlled study was used to ensure all participants received the intervention.

A content analysis was used to work with students as partners in the co creation of this intervention. To expand, students were asked about their views on immersive mindfulness, virtual reality, and procrastination, including suggestions on how they envisage the development of this intervention in supporting students. Student contributions included a whole person approach in co developing the intervention to target diverse students.

Virtual reality used Meta Quest 3 goggles with access to mindfulness software company. The intervention selected Focus mindfulness activities based on the impact of decision making, setting goals, being present, and working through barriers. Further, Calm was selected, focusing on flow, being in the here and now, and mindfully observing our senses and feelings with compassion. Post focus or calm, there was a series of mindfulness breathing exercises where participants could choose between the sea or land as a visual. A woman's voice provides guidance.

The mobile app uses artificial intelligence to provide personalised brief mindfulness exercises. Participants were encouraged to use this outside of virtual reality. The intervention has been mapped with mindfulness of breath, mindful stretching/body scan, mindful focus on difficulties and mindfulness of breath sounds and thoughts. Each session lasted approximately twenty five minutes per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have normal or corrected to normal hearing and vision
* Must be 8 years or older
* Must possess a mobile phone, either Google Play or Apple app
* Must have used virtual reality before with no side effects
* Must have a pulse rate of 60 to 80 beats per minute
* Must NOT experience seizures
* Must NOT have coordination difficulties

Exclusion Criteria:

* Have coordination difficulties
* Report having claustrophobia
* Pulse rate higher than 80 at rest
* Have sensitivities to flashing lights
* Are prone to migraine
* Have seizures
* Are younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Changes in cognitive mindfulness taken at weeks 0, 4 and 12 | 0, 4 and 12 weeks
  This is a 10 item questionnaire with 5 response categories (1=never or rarely true through 5=very often always true). Cronbach alpha ranges between 0.69 and 0.76. Subscale scoring is divided into 5 areas, including observing, describing, acting with awareness, non-judging, and non-reactivity. Higher scores reflect higher levels of mindfulness endorsement.
Changes in perceived academic stress taken at weeks 0, 4 and 12 | 0, 4 and 12 weeks
  This is a 10 item questionnaire with 5 response categories (1=Strongly disagree to 5=Strongly agree and in reverse 1= strongly agree to 5=strongly disagree). Cronbach alpha is .70. Primary subscales include academic expectations and self-perceptions. The higher the score, the higher the level of perceived academic stress experienced by students.
Changes in self efficacy taken at weeks 0, 4 and 12. | Weeks 0, 4 and 12
  This is a 15 item questionnaire with 5 response categories (1 = strongly disagree to 5 = strongly agree). Cronbach alpha is 0.85. The higher the score, the higher the level of self efficacy students experience.
Changes in academic engagement taken at weeks 0, 4 and 12 | Weeks 0, 4 and 12
  This is a 10 item questionnaire with 5 response categories (1 = strongly disagree to 5 = strongly agree). Cronbach alpha is 0.84. The higher the score the higher the level of academic engagement
Changes in academic procrastination taken at weeks 0, 4 and 12 | Weeks 0, 4 and 12
  This is a 10 item questionnaire with 5 response categories (1= disagree to 5= agree). It assesses procrastination in academic activities and settings. Cronbach alpha ranges between 0.84 and 0.92. The higher the score, the higher the level of perceived procrastination experienced by students.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Banbury, Principal Investigator — London Metropolitan University
Locations (1):
- School of Social Sciences and Professions, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boeldt D, McMahon E, McFaul M, Greenleaf W. Using Virtual Reality Exposure Therapy to Enhance Treatment of Anxiety Disorders: Identifying Areas of Clinical Adoption and Potential Obstacles. Front Psychiatry. 2019 Oct 25;10:773. doi: 10.3389/fpsyt.2019.00773. eCollection 2019. PMID 31708821
- [Result] Dundas I, Thorsheim T, Hjeltnes A, Binder PE. Mindfulness Based Stress Reduction for Academic Evaluation Anxiety: A Naturalistic Longitudinal Study. J College Stud Psychother. 2016 Apr 2;30(2):114-131. doi: 10.1080/87568225.2016.1140988. Epub 2016 Apr 13. PMID 27227169
- [Result] Biggers A, Spears CA, Sanders K, Ong J, Sharp LK, Gerber BS. Promoting Mindfulness in African American Communities. Mindfulness (N Y). 2020 Oct;11(10):2274-2282. doi: 10.1007/s12671-020-01480-w. Epub 2020 Aug 21. PMID 33584869
- [Result] Yue P, Zhang J, Jing Y. Mindfulness and academic procrastination among Chinese adolescents: a moderated mediation model. Front Psychol. 2024 Sep 2;15:1409472. doi: 10.3389/fpsyg.2024.1409472. eCollection 2024. PMID 39286568
- [Result] Koppenborg KA, Garnefski N, Kraaij V, Ly V. Academic stress, mindfulness-related skills and mental health in international university students. J Am Coll Health. 2024 Apr;72(3):787-795. doi: 10.1080/07448481.2022.2057193. Epub 2022 Apr 15. PMID 35427213
- [Result] Farra SL, Miller ET, Hodgson E. Virtual reality disaster training: translation to practice. Nurse Educ Pract. 2015 Jan;15(1):53-7. doi: 10.1016/j.nepr.2013.08.017. Epub 2013 Sep 12. PMID 24063793
- [Result] Ma J, Zhao D, Xu N, Yang J. The effectiveness of immersive virtual reality (VR) based mindfulness training on improvement mental-health in adults: A narrative systematic review. Explore (NY). 2023 May-Jun;19(3):310-318. doi: 10.1016/j.explore.2022.08.001. Epub 2022 Aug 5. PMID 36002363